CLINICAL TRIAL: NCT01638910
Title: A Multi-center, Open, Uncontrolled Phase 3 Study to Investigate the Efficacy and Safety of a 4-phasic Oral Contraceptive SH T00658ID Containing Estradiol Valerate and Dienogest in a 28-day Regimen for 13 Cycles in Healthy Female Subjects
Brief Title: Efficacy and Safety of a Combined Oral Contraceptive of Estradiol Valerate and Dienogest in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91773
Record Dates: First submitted 2012-06-20; First posted 2012-07-12 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Contraception
Keywords: Efficacy; Safety; oral contraception; estradiol valerate; dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EV/DNG (Qlaira, BAY86-5027) (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027) — Oral estradiol valerate and dienogest (2 days 3.0 mg estradiol valerate (EV), 5 days 2.0 mg EV + 2.0 mg dienogest (DNG), 17 days 2.0 mg EV + 3.0 mg DNG, 2 days 1.0 mg EV, 2 days placebo), one table oral daily for 13 treatment cycles (1 cycle = 28days)

SUMMARY:
To evaluate the efficacy and safety of a combined oral contraceptive of estradiol valerate and dienogest in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between 18 and 50 for the entire study, except women enrolled from India should be aged between 18 and 40 years, requesting contraception
* Smokers may not exceed 35 years of age

Exclusion Criteria:

* Pregnancy or lactation (delivery, abortion, or lactation within less than three cycles before the start of treatment)
* Body mass index (BMI) > 32 kg/m2
* Any disease or condition that may worsen under hormonal treatment
* Undiagnosed abnormal genital bleeding
* Other contraceptive methods such as sterilization, hormonal contraception, IUD within 30 days of Visit 1, monthly contraceptive injection within a period of three times of the injection interval before start of treatment
* Any medication that could result in excessive accumulation, impaired metabolism, or altered excretion of the study drug or interfere with the conduct of the study or the interpretation of the results

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 955 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of unintended pregnancies | Up to Cycle 13 (1 Cycle = 28 days)

SECONDARY OUTCOMES:
Number of expected bleeding days | Up to Cycle 13 (1 Cycle = 28 days)
Number of unexpected bleeding days | Up to Cycle 13 (1 Cycle = 28 days)
Number of expected bleeding episodes | Up to Cycle 13 (1 Cycle = 28 days)
Number of unexpected bleeding episodes | Up to Cycle 13 (1 Cycle = 28 days)
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Up to Cycle 13 (1 Cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (30):
- China (15):
  - Guangzhou, Guangdong
  - Shijiazhuang, Hebei
  - Wuhan, Hubei
  - Changsha, Hunan
  - Hengyang, Hunan
  - Nanjing, Jiangsu
  - Dalian, Liaoning
  - Shenyang, Liaoning
  - Jinan, Shandong
  - Chengdu, Sichuan
  - Wenzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Hong Kong, Hong Kong
- India (6):
  - Pune, Maharashtra
  - Chandigarh
  - Karnāl
  - New Delhi
  - Pune
  - Secunderabad
- Taiwan (5):
  - Taipei, Taipei
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok, Thailand
  - Bangkok
  - Chiang Mai

REFERENCES:
- [Derived] Yu Q, Huang Z, Ren M, Chang Q, Zhang Z, Parke S. Contraceptive efficacy and safety of estradiol valerate/dienogest in a healthy female population: a multicenter, open-label, uncontrolled Phase III study. Int J Womens Health. 2018 Jun 7;10:257-266. doi: 10.2147/IJWH.S157056. eCollection 2018. PMID 29922096